CLINICAL TRIAL: NCT02992158
Title: Feasibility of a Behavioral Activation Trial in Community Mental Health
Brief Title: Feasibility of a Behavioral Activation Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Merakey Behavioral Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH108818 (NIH)
Record Dates: First submitted 2016-12-01; First posted 2016-12-14 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2019-05

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- behavioral activation (Experimental): The core principles of the BA model are: (1) the key to changing how people feel is helping them change what they do, (2) changes in life can lead to depression, and short-term coping strategies may keep people stuck over time, (3) the clues to figuring out what will be antidepressant for a particular client lie in what precedes and follows the client's important behaviors, (4) structure and scheduling of activities should follow a plan, not a mood, (5) change will be easier when starting small, (6) activities that are naturally reinforcing should be emphasized, (7) the therapist should act as a coach, (8) a problem-solving empirical approach should be emphasized with recognition that all results are useful, (9) patients should be encourages to not just talk, do! (10) possible and actual barriers to activation should be examined. Patients can also receive medications in this arm.
  Interventions: Behavioral: behavioral activation
- treatment-as-usual (Other): Patients will receive psychotherapy (and potentially medications) as part of treatment-as-usual provided in the CMHC setting.
  Interventions: Behavioral: treatment-as-usual

INTERVENTIONS:
Behavioral: behavioral activation
  Arms: behavioral activation
Behavioral: treatment-as-usual — psychotherapy (and potentially medication) as part of treatment-as-usual provided in a community mental health center
  Arms: treatment-as-usual

SUMMARY:
The goal of this project is to train community mental health therapists in behavioral activation (BA) treatment for major depressive disorder and then to conduct a study examining the feasibility of evaluating the effectiveness of BA in this setting.

DETAILED DESCRIPTION:
After finalizing a 9-session BA treatment model for major depressive disorder in the Community Mental Health Center (CMHC) setting, the final treatment manual will be used to train clinicians in BA at the CMHC through workshops and training cases.

Upon completion of training and certification of adequate implementation of BA, a total of 80 patients with MDD will be randomly assigned in a 3:1 ratio to 9 sessions of BA or treatment-as-usual (TAU) at the CMHC. Feasibility will be assessed in terms of (1) percent of eligible patients who refuse randomization, (2) percent of patients who complete 9 sessions of BA treatment, (3) percent of BA homework assignments that are completed, (4) percent of monthly assessments obtained, and (5) patient ratings of credibility and alliance in BA treatment. The ability of CMHC therapists to adequately implement BA will be assessed by rating taped sessions on BA adherence and competence scales. In addition to feasibility/acceptability of BA and TAU, this study is designed to test whether theoretically important targets of BA change over the course of BA treatment, and whether such changes are associated with changes in depressive symptoms. The target measures will be assessed at baseline, month 1, month 2, and month 3. To support the potential role of these targets as the mechanisms of change in BA, change in the target variables will be examined in relation to change in depression symptoms. The investigators will also pilot a potential moderator of treatment effects (trait reward processing, as measured at baseline using the Effort-Expenditure for Rewards Task) to include this potential moderator in a subsequent fully-powered study with the long-term goal of identifying the types of patients most responsive to BA.

ELIGIBILITY:
Inclusion Criteria:

1. confirmed diagnosis of MDD based on the SCID for DSM-IV (or DSM-V, if available),
2. ability to read at least at the 4th grade level,
3. willingness to participate in research,
4. willingness to be audio recorded (for both therapists and patient- participants)

Exclusion Criteria:

1. current or past psychotic disorder, seizure disorder, or clinically significant organic pathology
2. acute medical problem requiring immediate inpatient treatment,
3. current substance abuse or dependence requiring primary referral to substance abuse program,
4. significant suicidal risk/ideation requiring immediate referral or suicidal gesture within the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
percent of eligible patients who refuse randomization | assessed at baseline
  We will calculate this value based on our records of patient participation in baseline assessments.
percent of patients who complete 9 sessions of BA treatment | 12 weeks
  We will calculate this value based on our records of patient attendance of therapy sessions (tracked each week by a research assistant).
percent of BA homework assignments that are completed | 12 weeks
  We will calculate this value based on our records of homework assignment completion (tracked weekly by therapist participants and reported to the research staff).
percent of monthly assessments obtained | 12 weeks
  We will calculate this value based on our records of patient assessment attendance (tracked by a research assistant).
Opinions About Treatment questionnaire | collected at week 2
  This questionnaire measures patient ratings of the credibility of BA treatment.
Brief Alliance Inventory | collected at weeks 2, 4, 6, and 8
  This questionnaire measures patient ratings of the therapeutic alliance.

SECONDARY OUTCOMES:
Behavioral Activation for Depression Scale | monthly for 3 months
Reward Probability Index | monthly for 3 months
Hamilton Rating Scale for Depression | monthly for 3 months
Short Form Health Survey (SF-36) | monthly for 3 months
Inventory of Depressive Symptomatology | monthly for 3 months
Behavior and Symptom Identification Scale (BASIS-24) | monthly for 3 months
Dysfunctional Attitudes Scale | monthly for 3 months
Quality of Life Index (questionnaire) | monthly for 3 months
Beck Anxiety Inventory | monthly for three months
Effort Expenditure for Rewards Task (EEfRT) | administered once at baseline and once at month 3

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared via the Research Domain Criteria Database (RDoCdb), part of the NIMH Data Archive (NDA). All feasibility and outcome data will be shared.